CLINICAL TRIAL: NCT06668038
Title: Evaluation of the Contribution of Multicenter Expertise (Radiotherapists and Physicists) and Use of Deformable Fusion Software Allowing the Accumulation of Doses in Equivalent Dose 2 Grays for Re-irradiations With Curative Intent
Brief Title: Contribution of Multicenter Expertise and Deformable Fusion Software for Re-irradiations With Curative Intent
Acronym: ADERE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADERE (ET23-390)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Re-irradiation; Radiotherapy
Keywords: Re-irradiation; Radiotherapy; Equivalent dose 2 grays; Feasibility; Cumulative doses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidisciplinary and multicenter validation of re-irradiation with curative intent (Experimental): Validation by a multicenter group of multi-professional experts (radiotherapists and physicists) of:
  * re-irradiation indication
  * EQD2 cumulated doses using MiM
  Interventions: Other: Multidisciplinary and multicenter validation of re-irradiation with curative intent

INTERVENTIONS:
Other: Multidisciplinary and multicenter validation of re-irradiation with curative intent — Validation in multidisciplinary and multicenter meeting of re-irradiation indication after review of technical data (images, structures and doses) of 1st irradiation and recent diagnosis images of the lesion to be irradiated, merged using MIM.
  In case of re-irradiation validation, validation in multidisciplinary and multicenter meeting of cumulated doses after review of EQD2 doses summation using MIM.

SUMMARY:
We propose to evaluate the contribution of a standardized process combining,

* a validation of re-irradiation indications by a group of multi-professional experts (radiotherapists and physicists) and,
* a collective validation of the accumulation of doses on all the organs of the anatomical region concerned obtained using deformable fusion software (MiM) allowing the accumulation of doses in terms of Equivalent Dose 2 Grays (EQD2).

The primary objective of this study is to determine the rate of patients for whom this process has changed the treatment plan.

DETAILED DESCRIPTION:
Recent clinical data confirm the possibility and clinical benefit of delivering a second irradiation with curative intent even if the commonly accepted maximum doses to OARs had been reached during the first irradiation.

However, there is no consensus on acceptable doses to AORs in a re-irradiation context. The difficulty of making decisions and validating dosimetry may limit access to treatment. Re-irradiations are therefore carried out according to local experience and equipment, resulting in territorial inequality.

MiM software is an innovative software dedicated to images registration and dose summation. It allows the EQD2 doses of the various irradiations to be cumulated.

Recruitment and inclusion step: For each included patient (signed consent form), the center provides an initial opinion concerning the indication for re-irradiation with curative intent (Opinion 1).

Indication and pre-dosimetric study step:

* If re-irradiation with curative intent Is not feasible according to the center: timages of the 1st irradiation and recent diagnosis images will be sent to Centre Léon Bérard (CLB), merged into MIM by physicists, and the indication is discussed in a multidisciplinary meeting (Opinion 2).
* If re-irradiation with curative intent is feasible according to the center: CT + RT structures+doses of 1st irradiation and dosimetric scan of the 2nd irradiation will be sent to CLB, merged into MIM. Multidisciplinary meeting will deliver the Opinion 3 with dosimetric instructions for the new irradiation, in particular OARs doses constraints.

Study withdrawal if the indication for re-irradiation is not validated.

Cumulative doses validation step:

CT + RT structures+doses of the planned re-irradiation will be sent to CLB and EQD2 doses will be summed into MIM. If cumulative doses are accepted by consensus, multidisciplinary meeting will deliver the Opinion 4. Otherwise the center will have to do a new planimetry.

Patients for whom re-irradiation with curative intent has been declared possible will be followed for 2 years according to standard practices, approximately every 3 months and analyzed for tolerance and efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years when signing the consent form
* Re-irradiation with desired curative intent (≥ 50 Gy EQD2), with volume to be irradiated totally or partially included in a previous irradiation field:

  * Oligo-metastases or oligo-progression (< 5 metastases in less than 3 sites)
  * Second non-metastatic cancer
  * Isolated local recurrence
* Life expectancy > 6 months
* Dated and signed informed consent
* Affiliation to a social security scheme or equivalent

Exclusion Criteria:

* Indication of intracranial, prostate, rectum or esophagus re-irradiation
* Diagnosis of multi-metastatic cancer
* PS ECOG ≥ 2
* Impossibility to interrupt current treatment with a tyrosine kinase inhibitor or other systemic treatment (excluding hormonal therapy) which may potentiate the rays effects (duration of wash-out according to treatment instructions)
* Pregnant or breastfeeding women
* Tutorship or curatorship or deprivation of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients for whom the intervention has changed the treatment plan | Up to 3 months
  Defined as the rate of patients for whom:
  * Re-irradiation at curative doses is finally possible while initially deemed unfeasible,
  * or validated median dose to GTV is increased by at least 5% compared to the initially envisaged dose,
  * or doses constraints to OARs are modified,
  * or the envisaged re-irradiation is invalidated.

SECONDARY OUTCOMES:
Late safety of re-irradiation | Up to 24 months
  Frequency of late (> 3 months after re-irradiation) grade ≥ 3 adverse events using NCI-CTCAE v5.0.
Local control rate at 3 months | At 3 months
  Rate of patients without progression in the field of re-irradiation
Local control rate at 6 months | At 6 months
  Rate of patients without progression in the field of re-irradiation
Local control rate at 12 months | At 12 months
  Rate of patients without progression in the field of re-irradiation
Local control rate at 24 months | At 24 months
  Rate of patients without progression in the field of re-irradiation
Time required for fusion and dose summation | Up to 3 months
  Median time for whole process workflow (fusion and dose summation)
Benefit of deformable registration | Up to 3 months
  Rate of patients with major anatomical changes between the 2 irradiations for whom the treatment plan was modified due to deformable registration compared to multiple rigid registrations carried out on different regions of interest
Rate of patients having received the proposed validated dose | Up to 5 months
  Rate of patients who received the re-irradiation dose as validated in multidisciplinary and multicenter meeting
Rate of patients without treatment-related toxicity or local progression or death at 2 years | Up to 24 months
  Number of patients without treatment-related toxicity ≥ 3 grade (according NCI-CTCAE v5.0) or local progression or death during the 2-year follow-up
Rate of change in centre practices | Up to 48 months
  Rate of centres in which re-irradiation practices have changed between study beginning and end.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre SUNYACH, Principal Investigator — Centre Leon Berard; Cécile LAUDE, Principal Investigator — Centre Leon Berard
Locations (10):
- France (10):
  - Institut de Cancerologie de L'Ouest, Angers
  - Ch Bourg En Bresse, Bourg-en-Bresse
  - Centre Georges Francois Leclerc, Dijon
  - Chu Grenoble Alpes, Grenoble
  - Centre Leon Berard, Lyon
  - Aphp Marseille Chu Timone Et Hopital Nord Marseille, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
  - Centre Marie Curie, Valence
  - Centre de Radiotherapie Du Beaujolais, Villefranche-sur-Saône